CLINICAL TRIAL: NCT03038451
Title: Efficacy and Safety of S-amlodipine 2,5 mg and 5 mg in Hypertension Patients: Open-label, Local, Phase IV Study
Brief Title: Efficacy and Safety of S-amlodipine 2,5 mg and 5 mg in Hypertension Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU-07.12
Record Dates: First submitted 2017-01-14; First posted 2017-01-31 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — levamlodipine; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- s-amlodipine besylate 2,5 and 5 mg tablets (Experimental)
  Interventions: Drug: S-NOR (s-amlodipine) 2,5 mg & 5 mg tablet

INTERVENTIONS:
Drug: S-NOR (s-amlodipine) 2,5 mg & 5 mg tablet

SUMMARY:
s-amlodipine besylate 2,5 mg tablet will be administered to patients have not received any hypertension treatment before or have received any of anti-hypertensive mono-therapy for the first four weeks of treatment. By increasing dose, s-amlodipine besylate 5 mg tablet will be administered for the last four weeks (4-8 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years and older.
* Hypertension patients have not received any anti-hypertensive treatment before ( ≥ 140 mmHg MSSBP < 160 mmHg, ≥ 90 mmHg MSDBP < 100mmHg).
* Hypertension patients controlled with single medicine.
* Patients giving written informed consent without being under any influence.

Exclusion Criteria:

* Pregnant patients, nursing mothers or female patients who have potential for childbearing and do not use any effective contraceptive method.
* Allergy or hypersensitivity to dihydropyridines.
* Patients receive more than one anti-hypertensive medicine.
* Patients with seconder hypertension.
* Patients with severe hypertension, myocardial infarction, NYHA stage 2-4 cardiac insufficiency, history of cerebrovascular disease, past ischemic attack, encephalopathy, underwent coronary artery bypass surgery or percutaneous coronary intervention, second or third degree heart block or symptomatic arrhythmia without pacemaker, clinically significant heart valve disease, potential life-threatening or symptomatic arrhythmia, simultaneous unstable angina pectoris, type I diabetes mellitus, atrial fibrillation until the last 12 months.
* Uncontrolled type II diabetes mellitus.
* Patients with significant liver disease (ALT, AST must be > 2XULN in beginning, patients with esophageal varices, portacaval shunt).
* Patients with significant kidney disease (GFR <60 ml/min according to Cockcroft-Gault formula).
* Patients with volume depletion.
* Patients with pancreas disease.
* Patients with gastrointestinal disease which may effect absorption.
* Drug/narcotic and alcohol abuse until the last 12 months.
* Patients with central nervous system disease and taking medicine for this reason.
* History of incompatibility with medical regimes or patients do not want to adhere the study protocol.
* Persons directly involved in the management of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2017-02-14 (Actual); Study Completion 2017-02-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of change in systolic blood pressure up to 4th week of the treatment | 4 weeks

SECONDARY OUTCOMES:
Evaluation of change in diastolic blood pressure up to 4th week of the treatment | 4 weeks
Evaluation of change in diastolic blood pressure up to 8th week of the treatment | 8 weeks
Evaluation of change in systolic blood pressure up to 8th week of the treatment | 8 weeks
Evaluation of change in systolic blood pressure from 4th to 8th week of the treatment | 4 to 8 weeks
Evaluation of change in diastolic blood pressure from 4th to 8th week of the treatment | 4 to 8 weeks
Evaluation of treatment response rates from 4th to 8th week of the treatment | 4 to 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University Istanbul Medical Faculty Clinical Pharmacology Department, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sen S, Demir M, Yigit Z, Uresin AY. Efficacy and Safety of S-Amlodipine 2.5 and 5 mg/d in Hypertensive Patients Who Were Treatment-Naive or Previously Received Antihypertensive Monotherapy. J Cardiovasc Pharmacol Ther. 2018 Jul;23(4):318-328. doi: 10.1177/1074248418769054. Epub 2018 Apr 12. PMID 29649885